CLINICAL TRIAL: NCT06516627
Title: Online Randomized Experiment Evaluating Front-of-Package Nutrition Labeling Systems
Brief Title: Front-of-Package Nutrition Labels
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard Pilgrim Health Care (Other)
Collaborators: Stanford University (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Jason Block, Associate Professor, Harvard Pilgrim Health Care
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1938853; R01DK115492 (NIH)
Record Dates: First submitted 2024-07-17; First posted 2024-07-24 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-08

CONDITIONS: Nutrition; Food Selection; Food Preferences; Dietary Habits; Healthy Diet
MeSH Terms: conditions — Food Preferences; Feeding Behavior | interventions — Product Labeling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Positive Labels (Experimental): Products that meet Guiding Stars' criteria for earning 1 or more Guiding Star will display labels indicating their healthfulness using star ratings: 1 star ("Good"), 2 stars ("Better"), or 3 stars ("Best"). The Guiding Stars rating system uses a patented algorithm to rate foods based on their nutrients and ingredients per 100-calorie serving of the food. Products that do not meet Guiding Stars' criteria for earning stars will not display any new front-of-package label.
  Interventions: Behavioral: Positive Labels
- Spectrum Labels (Experimental): All products will display an expanded Guiding Stars label that shows an overall rating indicating their healthfulness using star ratings: 1 star ("Poor"), 2 stars ("Fair"), 3 stars ("Good"), 4 stars ("Better"), or 5 stars ("Best"). The Guiding Stars rating system uses a patented algorithm to rate foods based on their nutrients and ingredients per 100-calorie serving of the food. Products that display 1-, 2-, or 3-star labels in the Positive Labels arm will display 3-, 4-, or 5-star labels, respectively, in the Spectrum Labels arm. The remaining products that do not earn stars in the Positive Labels arm will be divided in half based on their underlying Guiding Stars scores; the bottom half of these products will display 1-star labels and the top half of these products will display 2-star labels.
  Interventions: Behavioral: Spectrum Labels
- FDA High In Labels (Experimental): Products that contain high levels (i.e., ≥20% DV per serving) of saturated fat, sodium, or added sugars will display a label indicating which of these nutrients the product is high in. The investigators will use DVs of 20g for saturated fat, 2,300mg for sodium, and 50g for added sugars per FDA definitions.
  Interventions: Behavioral: FDA High In Labels
- FDA Traffic Light Labels (Experimental): All products will display a "Nutrition Info" label showing whether the amount of saturated fat, sodium, and added sugars in 1 serving of the product is low (<5% DV), medium (≥5 to <20% DV), or high (≥20% DV). "Low" will be shown in green, "Medium" in yellow, and "High" in red. The investigators will use DVs of 20g for saturated fat, 2,300mg for sodium, and 50g for added sugars per FDA definitions.
  Interventions: Behavioral: FDA Traffic Light Labels
- FDA High In Labels Plus Positive Labels (Experimental): Products that contain high levels (i.e., ≥20% DV per serving) of saturated fat, sodium, or added sugars will display a label indicating which of these nutrients the product is high in. The investigators will use DVs of 20g for saturated fat, 2,300mg for sodium, and 50g for added sugars per FDA definitions.
  Additionally, products that meet Guiding Stars' criteria for earning 1 or more Guiding Star will display labels indicating their healthfulness using star ratings: 1 star ("Good"), 2 stars ("Better"), or 3 stars ("Best"). The Guiding Stars rating system uses a patented algorithm to rate foods based on their nutrients and ingredients per 100-calorie serving of the food.
  Interventions: Behavioral: Positive Labels; Behavioral: FDA High In Labels
- FDA Traffic Light Labels Plus Positive Labels (Experimental): All products will display a "Nutrition Info" label showing whether the amount of saturated fat, sodium, and added sugars in 1 serving of the product is low (<5% DV), medium (≥5 to <20% DV), or high (≥20% DV). "Low" will be shown in green, "Medium" in yellow, and "High" in red. The investigators will use DVs of 20g for saturated fat, 2,300mg for sodium, and 50g for added sugars per FDA definitions.
  Additionally, products that meet Guiding Stars' criteria for earning 1 or more Guiding Star will display labels indicating their healthfulness using star ratings: 1 star ("Good"), 2 stars ("Better"), or 3 stars ("Best"). The Guiding Stars rating system uses a patented algorithm to rate foods based on their nutrients and ingredients per 100-calorie serving of the food.
  Interventions: Behavioral: Positive Labels; Behavioral: FDA Traffic Light Labels

INTERVENTIONS:
Behavioral: Positive Labels — Products that meet Guiding Stars' criteria for earning 1 or more Guiding Star will display labels indicating their healthfulness using star ratings: 1 star ("Good"), 2 stars ("Better"), or 3 stars ("Best").
  Arms: FDA High In Labels Plus Positive Labels; FDA Traffic Light Labels Plus Positive Labels; Positive Labels
Behavioral: Spectrum Labels — All products will display an expanded Guiding Stars label that show an overall rating indicating their healthfulness using star ratings: 1 star ("Poor"), 2 stars ("Fair"), 3 stars ("Good"), 4 stars ("Better"), or 5 stars ("Best").
  Arms: Spectrum Labels
Behavioral: FDA High In Labels — Products that contain high levels (i.e., ≥20% DV per serving) of saturated fat, sodium, or added sugars will display a label indicating which of these nutrients the product is high in.
  Arms: FDA High In Labels; FDA High In Labels Plus Positive Labels
Behavioral: FDA Traffic Light Labels — All products will display a "Nutrition Info" label showing whether the amount of saturated fat, sodium, and added sugars in 1 serving of the product is low (<5% DV), medium (≥5 to <20% DV), or high (≥20% DV). "Low" will be shown in green, "Medium" in yellow, and "High" in red.
  Arms: FDA Traffic Light Labels; FDA Traffic Light Labels Plus Positive Labels

SUMMARY:
The goal of this study is to determine whether certain front-of-package food labeling systems improve the healthfulness of consumers' grocery selections. US adults who are their households' primary shoppers will complete a shopping task in a naturalistic online grocery store. They will be exposed to different front-of-package food labeling systems and asked to shop for groceries. The online store will record participants' selections. Participants will also be asked to complete survey measures.

DETAILED DESCRIPTION:
This study aims to determine whether certain front-of-package food labeling systems improve the healthfulness of consumers' grocery selections. The survey research company Cloud Research will recruit a sample of approximately 5,610 US adults ages 18+ who read and speak English and who are their households' primary grocery shopper.

Participants will complete a between-subjects online randomized experiment. They will be randomized to 1 of 6 front-of-package labeling systems: 1) positive labels, 2) spectrum labels, 3) Food and Drug Administration (FDA) high in labels, 4) FDA traffic light labels, 5) FDA high in labels plus positive labels, or 6) FDA traffic light labels plus positive labels. Participants will complete a shopping task in a naturalistic online grocery store. Participants will be instructed to shop as they usually would for items in the following categories: non-alcoholic beverages (e.g., juice, coffee, tea, soda, sports drinks, water), breads and baked goods, breakfast cereals, soups, boxed and frozen meals, and snacks (e.g., chips, crackers, nuts, applesauce, dried fruit). They will be given a budget based on average spending in these categories in a large supermarket chain. The store will record participants' selections. After completing the shopping task, participants will complete an online survey.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older
* Reside in the US
* Can read and speak English
* Are their household's primary shopper (do 50% or more of the grocery shopping for their household)

Exclusion Criteria:

* Under the age of 18
* Reside outside of the United States
* Unable to complete a survey in English
* Are not their household's primary shopper (do <50% of the grocery shopping for their household)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5638 (Actual)
Dates: Start 2024-10-31 (Actual); Primary Completion 2024-11-21 (Actual); Study Completion 2024-11-21 (Actual)

PRIMARY OUTCOMES:
Healthfulness of participants' grocery selections | Assessed from enrollment to end of one-time, 30-minute online study survey
  The study will assess healthfulness of participants' grocery selections as the weighted average Ofcom Nutrient Profiling Model score of the products the participants select in the shopping task, weighted by the number of servings in each product. Ofcom Nutrient Profiling Model scores will be calculated for each product participants select. Products receive higher Ofcom scores when they contain lower calorie, saturated fat, sodium, and sugar density, higher protein and fiber density, and more fruits, vegetables, legumes, and nuts. The investigators will calculate the weighted average score across participants' selections, weighting by the number of servings participants select of that product. The Ofcom Nutrient Profiling Model score ranges from 0 to 100, where higher scores indicate healthier products.

SECONDARY OUTCOMES:
Guiding Stars scores of participants' grocery selections | Assessed from enrollment to end of one-time, 30-minute online study survey
  The study will assess Guiding Stars scores of participants' grocery selections as the weighted average Guiding Stars score of the products the participants select in the shopping task, weighted by the number of servings in each product. Products receive higher Guiding Stars scores when they contain more healthier nutrients and ingredients including vitamins, minerals, fiber, whole grains, and omega-3s and fewer unhealthy nutrients and ingredients including saturated fat, trans fat, added sodium, added sugars, and certain additives. Higher scores indicate healthier products.
Number of items selected that are high in ≥1 nutrient of concern | Assessed from enrollment to end of one-time, 30-minute online study survey
  The study will assess the number of items participants select that contain ≥20% DV of saturated fat, sodium, or added sugars. The investigators will use DVs of 20g for saturated fat, 2,300mg for sodium, and 50g for added sugars per FDA definitions. Higher counts will indicate a larger number of products selected were high in nutrients of concern.
Calorie density of participants' grocery selections | Assessed from enrollment to end of one-time, 30-minute online study survey
  The study will assess the weighted average calorie density of participants' grocery selections, calculated as the average kcal per 100g of the selected products, weighted by the number of servings in each product. Higher values will indicate higher calorie density.
Sugar density of participants' grocery selections | Assessed from enrollment to end of one-time, 30-minute online study survey
  The study will assess the weighted average sugar density of participants' grocery selections, calculated as the average grams of sugar per 100g of the selected products, weighted by the number of servings in each product. Higher values will indicate higher sugar density.
Sodium density of participants' grocery selections | Assessed from enrollment to end of one-time, 30-minute online study survey
  The study will assess the weighted average sodium density of participants' grocery selections, calculated as the average milligrams of sodium per 100g of the selected products, weighted by the number of servings in each product. Higher values will indicate higher sodium density.
Saturated fat density of participants' grocery selections | Assessed from enrollment to end of one-time, 30-minute online study survey
  The study will assess the weighted average saturated fat density of participants' grocery selections, calculated as the average grams of saturated fat per 100g of the selected products, weighted by the number of servings in each product. Higher values will indicate higher saturated fat density.
Fiber density of participants' grocery selections | Assessed from enrollment to end of one-time, 30-minute online study survey
  The study will assess the weighted average fiber density of participants' grocery selections, calculated as the average grams of fiber per 100g of the selected products, weighted by the number of servings in each product. Higher values will indicate fiber saturated fat density.
Protein density of participants' grocery selections | Assessed from enrollment to end of one-time, 30-minute online study survey
  The study will assess the weighted average protein density of participants' grocery selections, calculated as the average grams of protein per 100g of the selected products, weighted by the number of servings in each product. Higher values will indicate higher protein density.
Total calories selected | Assessed from enrollment to end of one-time, 30-minute online study survey
  The study will assess the total number of calories in participants' grocery selections, calculated as the sum of calories across all products selected. Higher values will indicate more calories selected.
Total sugar selected | Assessed from enrollment to end of one-time, 30-minute online study survey
  The study will assess the total amount of sugar in participants' grocery selections, calculated as the sum of sugar selected across all products selected. Higher values will indicate more sugar selected.
Total sodium selected | Assessed from enrollment to end of one-time, 30-minute online study survey
  The study will assess the total amount of sodium in participants' grocery selections, calculated as the sum of sodium selected across all products selected. Higher values will indicate more sodium selected.
Total saturated fat selected | Assessed from enrollment to end of one-time, 30-minute online study survey
  The study will assess the total amount of saturated fat in participants' grocery selections, calculated as the sum of saturated fat selected across all products selected. Higher values will indicate more saturated fat selected.
Total fiber selected | Assessed from enrollment to end of one-time, 30-minute online study survey
  The study will assess the total amount of fiber in participants' grocery selections, calculated as the sum of fiber selected across all products selected. Higher values will indicate more fiber selected.
Total protein selected | Assessed from enrollment to end of one-time, 30-minute online study survey
  The study will assess the total amount of protein in participants' grocery selections, calculated as the sum of protein selected across all products selected. Higher values will indicate more protein selected.
Total number of items selected | Assessed from enrollment to end of one-time, 30-minute online study survey
  The study will assess the total number of items participants select. Higher values will indicate more items selected.
Total spending on participants' grocery selections | Assessed from enrollment to end of one-time, 30-minute online study survey
  The study will assess the total amount participants spent on their grocery selections in USD. Higher values will indicate greater spending.
Correct identification of healthier items | Assessed from enrollment to end of one-time, 30-minute online study survey
  The study will assess the likelihood that participants correctly identify which of a pair of products is healthier with 6 items (1 for each of 6 product categories: bread, beverages, cereal, meals, snacks, and soups). Responses will be coded as correct (1) if participants select the product with the higher Ofcom Nutrient Profiling Model score and incorrect (0) otherwise.
Noticing of front-of-package labeling systems | Assessed from enrollment to end of one-time, 30-minute online study survey
  The study will assess noticing of the front-of-package labeling systems with 1 item: "When you were selecting foods and beverages in the shopping task, did you notice any other nutrition labels next to the products, besides the Nutrition Facts Panel?" Response options will be "yes," "no," and "not sure." Responses will be coded as noticed (1) if participants select "yes" and not noticed (0) otherwise.
Use of front-of-package labeling systems | Assessed from enrollment to end of one-time, 30-minute online study survey
  The study will assess use of the front-of-package labeling systems with 1 item: "While you were shopping, did you use these other nutrition labels to decide foods and beverages to select?" Response options will be "yes" (coded as 1) and "no" (coded as 0).
Thinking about health | Assessed from enrollment to end of one-time, 30-minute online study survey
  The study will assess thinking about health using 1 item: "When you were selecting foods and beverages in the shopping task, how much did you think about the overall healthfulness of the product? Response options range from not at all (1) to a great deal (5).
Negative emotional reactions | Assessed from enrollment to end of one-time, 30-minute online study survey
  The study will assess negative emotional reactions using 5 items: "How much does this label make you feel…" "worried", "scared," "guilty," "ashamed", and "sad"? Response options range from not at all (1) to a great deal (5). The investigators will average the 5 items; higher average scores indicate stronger negative emotional reactions.
Perceived helpfulness of the front-of-package labeling system | Assessed from enrollment to end of one-time, 30-minute online study survey
  The study will assess perceived helpfulness with 1 item: "How much do you agree or disagree with the following statement: These labels would help me choose healthier foods and beverages." Response options range from strongly disagree (1) to strongly agree (5).
Perceived understandability of the front-of-package labeling system | Assessed from enrollment to end of one-time, 30-minute online study survey
  The study will assess perceived understandability with 1 item: "How much do you agree or disagree with the following statement: It is easy to understand the information in these labels." Response options range from strongly disagree (1) to strongly agree (5).
Perceived trustworthiness of the front-of-package labeling system | Assessed from enrollment to end of one-time, 30-minute online study survey
  The study will assess perceived trustworthiness with 1 item: "How much do you trust or distrust the information in these labels?" Response options range from completely distrust (1) to completely trust (5).
Public support for front-of-package labeling system | Assessed from enrollment to end of one-time, 30-minute online study survey
  The study will assess public support for the front-of-package labeling systems with 1 item: "Would you oppose or support a policy requiring these labels on foods and beverages?" Response options range from strongly oppose (1) to strongly support (5).

CONTACTS AND LOCATIONS:
Overall Officials: Jason P. Block, MD, Principal Investigator — Harvard Pilgrim Health Care; Anna H. Grummon, PhD, Principal Investigator — Stanford University
Locations (1):
- Harvard Pilgrim Health Care Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Investigators will post de-identified individual participant data in a public repository.
Supporting Information: SAP, Analytic Code
Time Frame: Investigators will post IDP within 6 months of publication of manuscripts associated with the data generated in this study.
Access Criteria: Data and code will be made publicly available.

REFERENCES:
- [Derived] Huang Y, O'Sullivan K, Block JP, Petimar J, Lee CJY, Grummon AH. Impact of FDA's proposed front-of-package label and alternative designs on consumer understanding: A randomized experiment. Am J Prev Med. 2025 Dec 13:108222. doi: 10.1016/j.amepre.2025.108222. Online ahead of print. PMID 41397534
- [Derived] Grummon AH, O'Sullivan K, Petimar J, Lee CJY, Zeitlin AB, Cleveland LP, Collis C, Musicus AA, Tiefenbeck V, Fleisch E, Block JP. Nutrition Info and Other Front-of-Package Labels and Simulated Food and Beverage Purchases: A Randomized Clinical Trial. JAMA Netw Open. 2025 Oct 1;8(10):e2537389. doi: 10.1001/jamanetworkopen.2025.37389. PMID 41105412

DOCUMENTS (1):
  • Statistical Analysis Plan (2023-11-29): https://cdn.clinicaltrials.gov/large-docs/27/NCT06516627/SAP_000.pdf